CLINICAL TRIAL: NCT04397822
Title: Study of INFLAmmasome NLRP3 and PLAtelets Functions During Severe COVID-19 Infection
Brief Title: COVID-19 : Study of INFLAmmasome and PLAtelets Functions
Acronym: CO-QUETTES
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0142
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: COVID-19; NLRP3 inflammasome; Platelets functions; Coagulopathy; Acute respiratory distress syndrome
MeSH Terms: conditions — COVID-19; Hemostatic Disorders; Respiratory Distress Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 GROUP Intensive care unit: Patients suffering from COVID-19 hospitalized in intensive care unit
  Interventions: Biological: Blood samples
- COVID-19 GROUP Standard care unit: Patients suffering from COVID-19 hospitalized in standard care unit.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Blood samples will be collected in peripheral blood at the admission in intensive care unit or in standard care unit to compare platelet inflammasome NLRP3 and others markers

SUMMARY:
COVID-19 pandemic is a severe viral sepsis characterized by the occurrence of Acute respiratory distress syndrome (ARDS) whose pathophysiology is little described

DETAILED DESCRIPTION:
The new Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) epidemic started on December 2019 in China and spreaded in worldwide. The Coronavirus disease 2019 (COVID-19) is responsible of case of severe pneumonia whose the major risk is the development to ARDS. Concerning the pathophysiology, there appear to be hemostasis abnormalities including thrombocytopenia and coagulopathy. In recent studies, this thrombocytopenia is described as a risk factor to develop severe COVID-19 infection. Sepsis is associated with a major systemic inflammatory response with an increased production of pro-inflammatory cytokines. Since their discovery, inflammasomes have an important role during inflammatory response following an aggression. There are intracytoplasmic multiprotein complex activated by cellular stress or infections and is responsible for the release of pro-inflammatory cytokines, including IL-1β. Most studies have analysed inflammasomes in nucleated cells, nevertheless, little is known about inflammasomes in platelets.

Thus, the present work aims to study the activation of the platelet NLRP3 inflammasome and the platelet functions and coagulation during a SARS-CoV-2 viral pneumonia according to different levels of severity

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from COVID-19, hospitalized in intensive care unit and in standard care unit.

Exclusion Criteria:

* Patients suffering from malignant blood disease, cryopyrinopathy, sickle cell disease, rheumatoid arthritis and Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from COVID-19, hospitalized in intensive care unit and in standard care unit.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Activation of platelet NLRP3 inflammasome | Day 0 During resuscitation (Covid-19 Resuscitation) or hospitalization (Covid-19 No Resuscitation)
  Caspase-1 activity analyzed in patients in intensive care unit and in patients in standard care unit.
Activation of platelet NLRP3 inflammasome | During Day 0 During resuscitation (Covid-19 Resuscitation) or hospitalization (Covid-19 No Resuscitation)
  Labeling NOD-like receptor protein 3 (NLRP3)/Adaptor protein apoptosis-associated speck-like protein containing a CARD (ASC) analyzed in patients in intensive care unit and in patients in standard care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny BOUNES, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France